CLINICAL TRIAL: NCT06893016
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase 3 Study Evaluating the Safety, Tolerability, and Efficacy of RAY1225 in Participants Who Have Obesity or Are Overweight
Brief Title: Evaluation of RAY1225 in Adult Participants Who Have Obesity or Are Overweight
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Guangdong Raynovent Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RAY1225-24-07
Record Dates: First submitted 2025-03-18; First posted 2025-03-25 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- RAY1225 High Dose (Experimental): Participants will receive RAY1225 high dose subcutaneously (SC) for 52 weeks.
  Interventions: Drug: RAY1225
- RAY1225 Medium Dose (Experimental): Participants will receive RAY1225 Medium dose subcutaneously (SC) for 52 weeks.
  Interventions: Drug: RAY1225
- RAY1225 Low Dose (Experimental): Participants will receive RAY1225 low dose subcutaneously (SC) for 52 weeks.
  Interventions: Drug: RAY1225
- Placebo (Placebo Comparator): Participants will receive placebo SC for 52 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RAY1225 — RAY1225 will be administered SC
  Arms: RAY1225 High Dose; RAY1225 Low Dose; RAY1225 Medium Dose
Drug: Placebo — Placebo will be administered SC.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to demonstrate that RAY1225 is superior to placebo for percent change in body weight.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Body mass index ≥ 28 kg/m2 or ≥24kg/m² to <28 kg/m2 with at least 1 of the following weight-related comorbidities: a) Systolic blood pressure ≥130 mmHg or diastolic blood pressure ≥85 mmHg, or the use of at least one antihypertensive medication to maintain normal blood pressure;b) Fasting triglycerides (TG) ≥1.70 mmol/L, fasting low-density lipoprotein cholesterol (LDL-C) ≥4.1 mmol/L, fasting high-density lipoprotein cholesterol (HDL-C) <1.04 mmol/L, or the need for at least one lipid-lowering treatment to maintain normal lipid levels; c) Obstructive sleep apnea syndrome; d) Fatty liver; e) Cardiovascular disease; e) Polycystic ovary syndrome.
3. History of at least 1 self-reported unsuccessful attempt at weight loss by diet and exercise.

Exclusion Criteria:

1. Obesity known to be caused by monogenic mutations, other diseases, or medications.
2. Family or personal history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2.
3. A history of moderate to severe depression at any time in the past or a score of ≥15 on the PHQ-9 questionnaire at screening; a history of bipolar disorder, schizophrenia, or other severe psychiatric disorders.
4. A history of organ transplantation (excluding corneal transplant), or being currently prepared to undergo organ transplantation.
5. Plans to quit smoking during the study period
6. Allergic constitution (allergic to multiple medications or foods), or those known to be allergic to RAY1225, GLP-1 receptor agonists, or GLP-1 related drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Percent Change From Baseline in Body Weight at Week 52 | Baseline and Week 52
Number of Participants who Achieved a ≥ 5% Reduction in Body Weight from Baseline at Week 52 | Baseline and Week 52

SECONDARY OUTCOMES:
Change From Baseline in Waist Circumference at Week 52 | Baseline and Week 52

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided